CLINICAL TRIAL: NCT03790904
Title: Evaluation of Anti-plaque Effect of a Mouthwash Composed of Salvadora Persica L. and Green Tea: a 4days Randomized Controlled Crossover Clinical Trial
Brief Title: Anti Plaque Efficacy of Salvadora Persica L. and Green Tea Mouthwash
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hayder Raad Abdulbaqi, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 011618
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Periodontal Diseases
Keywords: Dental plaque,; Tea; Salvadora; Mouthwash; Clinical trial
MeSH Terms: conditions — Periodontal Diseases; Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co. mouthwash (Active Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Co.
- Kin mouthwash (Placebo Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Kin
- Distilled water (Placebo Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Distilled water

INTERVENTIONS:
Other: Co. — 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: Co. mouthwash
Other: Kin — 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: Kin mouthwash
Other: Distilled water — 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: Distilled water

SUMMARY:
Periodontal diseases and caries are essentially initiated and progressed by accumulation of dental plaque. Thus, daily effective plaque control is valuable as a preventive measure and maintaining oral health. Mechanical plaque control is important but has limitations; therefore, an adjunctive chemical plaque control such as mouthwash is helpful. Various medicinal plant-derived galenicals might be used as safe and stable alternatives to synthetic mouthwashes. For example, a combination of Salvadora persica L. (Sp) root sticks and green tea (Gt) aqueous extract has been found to reduce plaque accumulation over 24 hours. Moreover, these extracts were reported to have anti-microbial activity against many oral bacteria. The objective of this study was to investigate the efficacy of the combination of Gt aqueous extract and Sp aqueous extract in reducing plaque buildup for 4 days duration.

DETAILED DESCRIPTION:
Dental plaque is the soft mass formed on oral surfaces including tooth surfaces. It composed of many species of which are commensal and other are pathogenic. The buildup of dental plaque starts by adhesion of floating bacteria, primary colonizers, in saliva onto oral surfaces such as tooth surfaces. Consequently, after adhesion, these primary bacteria provide adhesion sites for secondary plaque colonizers and the plaque buildup continues to achieve a mature dental plaque.

The mature dental plaque initiates host immune response by its bacterial content or its toxins in the adjacent gingival tissues. Periodontal health is assumed to be in a state of balance when the host immune response resolves the bacterial challenges. In other scenario, the host immune response fails to overcome invader bacteria or their toxins leading to chronicity of aberrant immune responses. Thus, periodontal diseases and caries may be developed due to imbalance between dental plaque accumulation and host defense. For that reason, dental plaque control is essential as preventive measure for good oral health.

Mechanical plaque control including tooth brushing and interdental aids is essential for preserving oral health. However, efficient mechanical control is time consuming and needs high manual dexterity and compliance. Therefore, chemical plaque control such as mouthwashes might be useful as adjunctive to mechanical control. Chlorohexidine mouthwash is the best-known mouthwash serving that purpose despite its side effects including tooth discoloration and bitter taste.

Salvadora persica L. (Sp) root sticks and green tea (Gt), leafs of Camellia sinensis, aqueous extracts were reported to exert anti-microbial activity against many oral bacteria. A combination (Co.) of Gt aqueous extract and Sp aqueous extract at a specific concentration (patented, IP 2015704777) was found to exhibit significant synergistic anti-bacterial and anti-adherence efficacy against primary plaque colonizers in vitro. This Co. as a mouthwash was reported to significantly reduce plaque accumulation comparing to chlorhexidine in vivo for a period of 24 hours (NCT02624336 in December 3, 2015).

ELIGIBILITY:
Inclusion Criteria:

* Participants should be medically healthy.
* Participants should have more than 20 teeth.

Exclusion Criteria:

* Participants who have active cavity caries and/or periodontal disease.
* Participants who have ongoing orthodontic treatment.
* Participants who have been on antibiotics within the past 4 months.
* Participants who require prophylactic antibiotic coverage.
* Participants who have been on systemic or topical non-steroidal anti-inflammatory drugs for the past 4 months.
* Participants who are pregnant or intended to and lactating mother.
* Participants who have heart valve replacement and have known intolerance or allergy to mouth rinses.
* Participants who have any systemic disease.

Ages: 20 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Mean amount plaque between different comparators | Time Frame: 24 hours
  Mean amount plaque between different comparators as anti-plaque agent following 24 hrs plaque regrowth clinical trial by means of modified quigely hein plaque index [Turesky, 1970] and digital plaque image analysis.
Mean amount plaque between different comparators | Time Frame: 4 days
  Mean amount plaque between different comparators as anti-plaque agent following 4 days plaque regrowth clinical trial by means of modified quigely hein plaque index [Turesky, 1970] and digital plaque image analysis.

SECONDARY OUTCOMES:
Mean bacterial load in saliva | 2 hours
  Mean bacterial load in saliva at 2 hours after rinsing with different comparators using quantitative polymerase chain reaction (qPCR).
Mean relative changes in gingival crevicular fluid flow rate | 4 days
  Mean relative changes in gingival crevicular fluid flow rate after rinsing with different comparators from baseline at 4 days.
Mean relative changes in Interleukin1 beta levels in gingival crevicular fluid | 4 days
  Mean relative changes in Interleukin1 beta levels in gingival crevicular fluid after rinsing with different comparators from baseline at 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha S Abbood, Principal Investigator — University of Baghdad
Locations (1):
- Hayder R Abdulbaqi, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided